CLINICAL TRIAL: NCT02282150
Title: Effect of Modified-release Compared to Conventional Hydrocortisone on Fatigue, Measured by Ecological Momentary Assessments; a Pilot Study.
Brief Title: Modified-release Compared to Conventional Hydrocortisone on Diurnal Fatigue in Secondary Hypoadrenalism
Acronym: PlenadrEMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ulla Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Ulla Feldt-Rasmussen, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLEN-EMA-hypo; 2014-002039-32 (EudraCT Number); H-1-2014-073 (Other: Health Research Ethics in Capital Region of Denmark)
Record Dates: First submitted 2014-10-26; First posted 2014-11-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Adrenal Insufficiency
Keywords: Fatigue; Quality of Life; Hydrocortisone; Ecological Momentary Assessments
MeSH Terms: conditions — Adrenal Insufficiency; Fatigue | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Cross over
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conventional vs modified hydrocortisone; (Other): 5 weeks of conventional hydrocortisone followed by 16 weeks of modified-release hydrocortisone (Plenadren)
  Interventions: Drug: Hydrocortisone; Drug: Plenadren

INTERVENTIONS:
Drug: Hydrocortisone — Usual hydrocortisone dosage regimen; 10-40 mg hydrocortisone administered twice or thrice daily for 5 weeks
Drug: Plenadren — 10-40 mg modified-release hydrocortisone in tablets, once a day for 16 weeks
  Other Names: Modified-release hydrocortisone

SUMMARY:
Despite optimized hydrocortisone replacement regimes, many patients with adrenal insufficiency (AI) suffer from impaired quality of life (QoL). Characteristically, patients report high fatigue levels at certain times during the day. A modified-release hydrocortisone has been shown to improve QoL, particularly fatigue, in patients with primary AI. However, it is unknown, if the same effect can be observed in patients with secondary AI. Further, no studies have evaluated the effect, taking into account the diurnal variation of fatigue. A novel survey method termed Ecological Momentary Assessments (EMA) has the potential to provide reliable measurements of diurnal variations in patient-reported outcomes, such as fatigue. We will compare the effect of modified-release compared to conventional hydrocortisone on fatigue in patients with secondary AI due to pituitary disease, and hereby assess the feasibility of EMA as outcome in future large-scale randomised clinical trials (RCTs).

DETAILED DESCRIPTION:
The study is conducted as an open-label, single-arm, two-period, crossover pilot trial. Includible patients are observed for 5 weeks on their usual treatment (twice or thrice daily hydrocortisone). Assessments of QoL, in terms of EMA assessments, to be used as baseline measurement in the study, are collected for 20 days preceded by a 5 days technology adaptation phase. Thereafter participants are shifted to modified release hydrocortisone (Plenadren) once daily (OD), on a dose as per Summary of Product Characteristics (SmPC). Assessments of QoL to be used as outcome of intervention in the study are performed after 12.5 weeks after initiation of Plenadren intervention treatment, in order to take into consideration the period of re-adjustment of the body after the switch from conventional hydrocortisone to Plenadren. As done at the baseline observation, EMA measurement is preceded by a five days technology adaptation phase. At the end of the intervention treatment period, the patients will be shifted to their usual hydrocortisone treatment and will be followed at the outpatient clinic according to the directives of the clinic. Biochemical parameters; blood samples, DEXA scan, 24 hour blood pressure and salivary cortisol, will be assessed at baseline and after 16 weeks, as part of the safety evaluation of Plenadren.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adrenal insufficiency due to hypopituitarism
* In steady twice or thrice daily (10-40 mg) hydrocortisone replacement treatment
* Written informed consent
* For women: Use of reliable methods of contraception in clinical trials in accordance with the definition by the Danish Health and Medicines Authority; intrauterine devices or hormonal methods (oral contraceptives, contraceptive implants, transdermal patches, hormonal vaginal devices or injections with prolonged release).

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Acromegaly
* Cushing's Disease
* Diabetes Mellitus
* Other major confounding disease
* Known or expected hypersensitivity to any of the excipients
* Lack of compliance (attendance and medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment (EMA) fatigue profiles | 25 days during conventional hydrocortisone treatment and for 25 days during Plenadren (intervention) treatment
  Differences and variability of standard treatment vs. modified release hydrocortisone EMA fatigue profiles

SECONDARY OUTCOMES:
Quality of Life questionnaires | At baseline and after 16 weeks of Plenadren (intervention) treatment
  Fatigue Impact Scale (FIS), AD-specific quality-of-life questionnaire (AddiQol) and the Short Form Health Survey (SF-36)
Safety (Biochemical parameters, DEXA scan, 24 hour blood pressure and salivary cortisol) | At baseline and after 16 weeks of Plenadren (intervention) treatment
  Biochemical parameters, DEXA scan, 24 hour blood pressure and salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: Undecided